CLINICAL TRIAL: NCT02510196
Title: Assessment of Skill Retention in Clinical Practice
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 0036-13-HMO
Record Dates: First submitted 2015-06-10; First posted 2015-07-29 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2015-02

CONDITIONS: Risk Reduction
MeSH Terms: conditions — Risk Reduction Behavior

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- reminder (Active Comparator): participants in this group will be reminded to use ultrasound for neuraxial anesthesia on a regular basis
  Interventions: Behavioral: reminder
- control (No Intervention): participants in this group will not be reminded to use ultrasound for neuraxial anesthesia

INTERVENTIONS:
Behavioral: reminder
  Arms: reminder

SUMMARY:
Teaching program population: Participants in Hadassah Ein Kerem ultrasound training day - Anesthesia residents Exclusion criteria: Refusal to participate, insufficient understanding of written English used in the questionnaires

Stage 1 - training The aims and requirements of the teaching program will be explained to the participants at the start of the workshop. All participants will be given a sticker with a number and a questionnaire numbered about current ultrasound practice which is numbered according to participant number to allow for blinding. Anyone not wishing to participate can either remove their sticker or not return the questionnaire at the end of the session. The number on the questionnaire correlated to participant number. This will be recorded against the participant name to allow for further follow up. All participants will rotate normally throughout the sessions. At the end of the neuraxial session participants will be scored by the session leader according to their ability to adequately carry out the procedure. Scores will be correlated to participant number.

Stage 2 - assessment of skill retention

Following the training day participants will randomly be allocated into two groups. One group will receive regular reminders to use ultrasound for all neuraxial anesthesias they perform in the OR or labor ward. They will be reminded on a regular basis that ultrasound is a new tool to assist them in performing neuraxial ultrasound. The other group with be allowed to continue with their regular practice and will not receive reminders to use ultrasound for neuraxial anesthesia insertion. Two months after the initial training day all participants with be observed performing neuraxial anesthesia and re-assesed according to the original scoring system. Each participant will be assessed 3 times over a 6 month period.

ELIGIBILITY:
Inclusion Criteria:

* Practicing anesthesiologists of all levels at Hadassah Ein Kerem hospital

Exclusion Criteria:

* Unwillingness to complete questionnaire, poor English comprehension

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-04; Primary Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Ultrasound Performance on a model | 1 year
  ability of participants to perform neuraxial ultrasound will be assessed at 2 monthly intervals